CLINICAL TRIAL: NCT04967560
Title: The Efficacy and Safety of Deep Brain Stimulation of Combined Anterior Limb of Internal Capsule and Nucleus Accumbens (ALIC/NAcc-DBS) for Treatment-refractory Obsessive-compulsive Disorder (OCD)
Brief Title: The Efficacy and Safety of ALIC/NAcc-DBS for Treatment-refractory OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: West China Hospital (Other); Huashan Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Hunan Brain Hospital (Unknown); First Affiliated Hospital of Kunming Medical University (Other); Changhai Hospital (Other); SceneRay Corporation, Limited (Industry)
Responsible Party: Principal Investigator, Zhen Wang, Shanghai Mental Health Center, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SR1182
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: obsessive-compulsive disorder; deep brain stimulation; anterior limb of internal capsule; nucleus accumbens
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: All eligible patients who consent to participation and met all inclusion and exclusion criteria will be randomized to active and sham-stimulation group at post-operative.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization of DBS are blinded to evaluators, participants, and programming doctors. The programming doctors used the specific software to allocated the participants, that software was preset random coding program to randomized allocate the subjects. The DBS interface of all patients is displayed as a true stimulus, but the true impulse was running in the background controlled by the software, so that even the programming doctors could not know the grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DBS true-stimulation group (Active Comparator): The electrical stimulation will be 'turned-on' immediately after programming in true-stimulation group.
  Interventions: Device: deep brain stimulation
- DBS sham-stimulation group (Sham Comparator): The electrical stimulation will be 'turned-off' after programming in sham-stimulation group. The stimulation will begin until after completing three months of Y-BOCS and CGI assessments
  Interventions: Device: deep brain stimulation

INTERVENTIONS:
Device: deep brain stimulation — Both group will undergo the DBS surgery. Four weeks after surgery, all patients will visit the clinic with the DBS stimulation in the 'off' state for initial programming of electrical parameters for stimulation. At double-blind visit, the electrical stimulation will be actually 'turned on' immediately after the programming in true-stimulation group, while turn-off in the control group.

SUMMARY:
The present study aims to explore the efficacy and safety of DBS targeted the combination of the anterior limb of internal capsule and nucleus accumbens (ALIC/NAcc-DBS) to refractory OCD, based on multicenter, randomized, double-blinded, sham-stimulation controlled design, that could help to obtain stronger evidence of the efficacy of multiple targets.

DETAILED DESCRIPTION:
OCD is a chronic and disabled mental disorder, with one third of patients could hardly get recovery from the medication and psychotherapy. Deep brain stimulation (DBS) is a novel potential surgical treatment for refractory OCD, however, the choose of targets are still controversial. This study aims to investigate the therapeutic efficacy and safety of bilateral DBS of the anterior limb of internal capsule and nucleus accumbens (ALIC/NAcc-DBS) for treatment-refractory OCD. In this multicenter, prospective, and double-blinded study, 64 patients with OCD who met the eligibility criteria will be enrolled and randomized allocated to active and sham-stimulation group, followed up for three months after surgery. Then the blind will be uncover, the sham group switch to true stimulation, all patients will be followed up at six months after surgery. The primary outcome was to compare the treatment response rate between the active group and sham-controlled group at the end of three months after surgery. The secondary outcomes include changes in the Yale-brown obsessive-compulsive scale (Y-BOCS), Hamilton anxiety scale (HAMA), Hamilton depression scale (HAMD), and Clinical global impressions (CGI) scale of both groups.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years old;
* a diagnosis of OCD based on The Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5);
* suffered from severe OCD symptoms over 5 years with substantial functional impairment;
* the Y-BOCS total score ≥ 25;
* met the criteria of treatment refractory. Treatment refractory is defined as failed 1) at least three adequate therapeutic trials of serotin reuptake inhibitors (SRIs), with clomipramine being one of the SRIs trials, 2) the use of at least two atypical antipsychotics as augmenting agents, 3) at least 20 sessions of therapist-guided cognitive-behavioral therapy while on a therapeutic dose of an SRIs. These patients have "failed" treatment by demonstrating <25% reduction of Y-BOCS scores or, despite >25% reduction in YBOCS score, by still experiencing significant impairment from their illness.

Exclusion Criteria:

* a history of current or past diagnosis of any psychosis according to DSM-5 except for OCD
* any clinical significant neurological disorder, traumatic brain injury, dementia, or medical illness
* any contradiction of neurosurgery
* any current or unstably remitted substance abuse or dependence
* women who are pregnant or preparing for pregnant
* severe suicide risk and tendency according to the investigators' judgements
* participate in any other clinical trials within three months (except for registered studies).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Treatment response rate | three month after stimulus
  Our primary outcome measure was to compare the treatment response rate (TRR) between the active group and sham-controlled group at the end of three months. (TRR is defined as the number of treatment response/the number of group, a ≥35% reduction in Y-BOCS plus CGI=1or2 met the criteria of treatment response). Note: Y-BOCS, Yale-Brown obsessive-compulsive scale; CGI, clinical global impression.

SECONDARY OUTCOMES:
the change scores of Y-BOCS at double-blinded stage | three month after stimulus
  The severity of OCD symptoms was assessed using the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS). This scale including 10 items, the maximum score is 40. The higher score means the more serious of disease.
the change scores of CGI at double-blinded stage | three month after stimulus
  The Clinical Global Impressions (CGI) is an invaluable tool for monitoring the treatment outcomes of patients.The CGI actually comprises three companion one-item measures evaluating the following: (a) severity of psychopathology from 1 to 7, (b) change from the initiation of treatment on a similar seven-point scale, and (c) an overall evaluation of the theraputic effect and side effects.
the change scores of HAMD at double-blinded stage | three month after stimulus
  The Hamilton Depression Rating Scale (HAM-D) is used to quantify the severity of symptoms of depression and is one of the most widely used and accepted instruments for assessing depression. It contains 24 items rated on 5-point scale, with the sum of all items making up the total score, yielding total scores from zero to 96. The higher score means more severity of depression symptoms.
the change scores of HAMA at double-blinded stage | three month after stimulus
  The Hamilton Anxity Rating Scale (HAM-A) was one of the first rating scales developed to measure the severity of anxiety symptoms. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety and somatic anxiety. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
the change scores of Y-BOCS at open-label stage | six month after stimulus
  The severity of OCD symptoms was assessed using the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS). This scale including 10 items, the maximum score is 40. The higher score means the more serious of disease.
the change scores of CGI at open-label stage | six month after stimulus
  The Clinical Global Impressions (CGI) is an invaluable tool for monitoring the treatment outcomes of patients.The CGI actually comprises three companion one-item measures evaluating the following: (a) severity of psychopathology from 1 to 7, (b) change from the initiation of treatment on a similar seven-point scale, and (c) an overall evaluation of the theraputic effect and side effects.
the change scores of HAMD at open-label stage | six month after stimulus
  The Hamilton Depression Rating Scale (HAM-D) is used to quantify the severity of symptoms of depression and is one of the most widely used and accepted instruments for assessing depression. It contains 24 items rated on 5-point scale, with the sum of all items making up the total score, yielding total scores from zero to 96. The higher score means more severity of depression symptoms.
the change scores of HAMA at open-label stage | six month after stimulus
  The Hamilton Anxity Rating Scale (HAM-A) was one of the first rating scales developed to measure the severity of anxiety symptoms. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety and somatic anxiety. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Brains Hospital of Hunan Province, Changsha, Hunan
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No